CLINICAL TRIAL: NCT05608369
Title: A Phase 2 Study of Vorinostat in Combination With Chemoradiation in Patients With Locally Advanced HPV Negative HNSCC
Brief Title: Vorinostat in Combination With Chemoradiation in Locally Advanced HPV Negative HNSCC
Acronym: HPV
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2321
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: HPV-Related Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Oral Cavity; Squamous Cell Carcinoma of the Larynx; Squamous Cell Carcinoma of the Oropharynx; Squamous Cell Carcinoma of the Hypopharynx
Keywords: Squamous Cell Carcinoma; HPV-Related Squamous Cell Carcinoma; Chemoradiation; Locally Advanced HPV negative HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — Cisplatin; Radiotherapy; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study drug + Standard of care chemoradiation (Experimental): Participant will be pre-treated with study drug followed by continuation of standard chemoradiation
  Interventions: Drug: Cisplatin; Radiation: Radiation therapy; Drug: Vorinostat

INTERVENTIONS:
Drug: Cisplatin — Cisplatin100 mg/m2 every 3 weeks or 40 mg/m2 weekly
Radiation: Radiation therapy — Radiation therapy (70 Gy) for total of 7 weeks
Drug: Vorinostat — Pre-treatment; 300 mg every other day and ends with the dose closest to the last fraction of radiation (total of 8 weeks)

SUMMARY:
The purpose of this study is to learn more about a drug called Vorinostat (an experimental drug) in combination with chemoradiation. The intention of this study is to learn if this drug is safe for the participants and whether this drug with chemoradiation is able to further increase the clinical efficacy of chemoradiation, which is an approved therapy. The main question it aims to answer is: How may Vorinostat interact with standard chemotherapy and radiation therapy in head and neck cancer? Participants will receive the study drug (Vorinostat) as a pre-treatment, followed by standard chemoradiation.

DETAILED DESCRIPTION:
Histone deacetylase (HDAC) inhibitors have been shown to increase reverse resistance to cisplatin and radiation therapy. This phase 2 study comes after an already completed phase 1 study which examined tolerability of pan-HDAC inhibitor, Vorinostat, in combination with chemoradiation in locally advanced head and neck squamous cell carcinoma (HNSCC). The study showed that Vorinostat in combination with concurrent chemoradiation therapy (CRT) is safe and estimated 5-year OS of HPV- patients is 77.8% which is considerably higher than the 5-year overall survival (OS) of 46.2% in HPV- HNSCC patients treated with standard concurrent chemoradiation. Based on this phase 1 study, the hypothesis is that Vorinostat, in combination with chemoradiation, will increase median progression-free survival compared to chemoradiation alone treatment in HPV-HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed stage III or IV HPV negative squamous cell carcinoma of the oral cavity, oropharynx or hypopharynx, tumors is deemed to be either unresectable or locally advanced.
* Subjects must have received no prior therapies (chemotherapy or radiotherapy) for this disease
* Age >18 years. Because the low occurrence of HNSCC in the pediatric population, children are excluded from this study
* ECOG Performance status ≤ 2
* Subjects must have normal organ and marrow function as defined below

  * Hemoglobin ≥ 9.0 g/dl (transfusion permitted)
  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 100,000/mcL
  * Total bilirubin within normal institutional limits
  * AST (SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Serum Creatinine clearance (> 50 ml/min)
* Based on findings from animal studies and its mechanism of action, vorinostat can cause fetal harm when administered to a pregnant woman. There are insufficient data on vorinostat use in pregnant women to inform a drug-associated risk of major birth defects and miscarriage. In animal reproduction studies, vorinostat crossed the placenta and caused adverse developmental outcomes at exposures approximately 0.5 times the human exposure based on AUC0-24 hours. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) beginning at study entry and for the duration of study participation. Male study participants should use an additional barrier method of contraception for 30 days following the last dose of vorinostat. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Patients must have measurable disease, per RECIST 1.1
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Eligibility for curative-intent surgery, previous chemotherapy.
* Subjects receiving any other investigational agents.
* Subjects with untreated brain metastases/CNS disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat.
* Patients with previous exposure to vorinostat.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because vorinostat may have potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with vorinostat, breastfeeding should be discontinued if the mother is treated with vorinostat. These potential risks may also apply to other agents used in this study.
* HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with vorinostat. In addition, these subjects are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in subjects receiving combination antiretroviral therapy when indicated. Also include whether HIV testing is required for this study, or only if a known diagnosis will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Through completion of follow-up (estimated to be 2.5 years)
  Determine progression free survival (PFS) of patient with locally advanced HPV- HNSCC treated with vorinostat and standard chemoradiation (CRT).

SECONDARY OUTCOMES:
Objective response rate | Through completion of follow-up (estimated to be 2.5 years)
  Determine objective response rate (ORR), overall survival (OS) of patient with locally advanced HPV- HNSCC treated with vorinostat and standard chemoradiation (CRT).

CONTACTS AND LOCATIONS:
Overall Officials: Kyunghee Burkitt, DO, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie or influence the results observed in this study
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Investigators who provide a methodologically sound proposal for use of requested data